CLINICAL TRIAL: NCT00879073
Title: Phase I Study of Bendamustine With Concurrent Whole Brain Radiation Therapy in Patients With Brain Metastases From Solid Tumors
Brief Title: Study Bendamustine Concurrent Whole Brain Radiation Brain Metastases From Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator is leaving Moffitt
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network); Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15690
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Brain Metastases
Keywords: Brain and Nervous System
MeSH Terms: conditions — Brain Neoplasms; Neurologic Manifestations | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A - Cohort 1 Treatment (Experimental): Cohort 1: Bendamustine 60 mg/m² x 4 weeks
  Interventions: Drug: Bendamustine
- B - Cohort 2 Treatment (Experimental): Cohort 2: Bendamustine 80 mg/m² x 4 weeks
  Interventions: Drug: Bendamustine
- C - Cohort 3 Treatment (Experimental): Cohort 3: Bendamustine 100 mg/m² x 4 weeks
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — Approximately 15-24 study patients will be enrolled in this Phase I trial. Study patients will receive a weekly dose of IV bendamustine with whole brain radiation therapy for 3 weeks and then receive a fourth dose of IV bendamustine one week after completion of whole brain radiation therapy. The first dose of IV bendamustine will be given when whole brain radiation is initiated.
  Other Names: Treanda

SUMMARY:
The purpose of this study is to:

* Test the maximum tolerated dose (MTD) of Bendamustine with whole brain radiation therapy (WBRT)
* To determine the plasma pharmacokinetics (a blood test to see how much of the drug is getting into the patient's system and how long it lasts in the system) of Bendamustine
* To determine the presence of Bendamustine in cerebrospinal fluid (CSF) (fluid from the brain and spinal cord) of study patients Bendamustine is approved by the Food and Drug Administration (FDA) for chronic lymphocytic leukemia. However, Bendamustine will be used in this study as an investigational agent.

DETAILED DESCRIPTION:
Bendamustine will be started in the first group at a dose of 60 mg/m²; patients in group 2 will be given Bendamustine at a dose of 80 mg/m²; patients in Group 3 will be given Bendamustine at 100 mg/m². Each cohort will receive Bendamustine once weekly for a total of 4 weeks.

Approximately 3-6 patients enrolled in this study will receive lumbar punctures. Patients will be told before study enrollment whether they will have a lumbar puncture to withdraw CSF.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of solid tumor malignancy within 5 years of registration. Pathological confirmation by pathologists at Moffitt Cancer Center is required.
* Cerebral metastases from known solid tumors diagnosed by contrast-enhanced brain magnetic resonance imaging (MRI) or contrast-enhanced head computed tomography (CT) for patients unable to receive MRIs
* Single metastases that have been resected
* Patient may have had prior radiosurgery or surgical resection for brain metastasis. Patients should have completed prior therapy at least 14 days but no longer than 56 days prior to study entry.
* Karnofsky Performance Status ≥ 70 within 28 days prior to study entry.
* Expected life span of ≥ 3 months
* Able to tolerate 3 week course of whole brain radiation therapy
* Able to receive a lumbar puncture (for post-MTD patients only)
* Adequate bone marrow, liver and renal function as assessed by the following: Hemoglobin > 9.0 g/dl; Absolute neutrophil count (ANC) > 1,500/mm³; Platelet count > 100,000/mm³; Total bilirubin < 1.5 x upper limit of normal (ULN); Alanine transaminase/Aspartic transaminase (ALT/AST) < 2.5 x the ULN (< 5 x ULN for patients with liver involvement); International normalized ratio (INR) < 1.5 or a prothrombin time/partial thromboplastin time (PT/PTT) within normal limits; Creatinine < 1.5 x ULN
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Ability to understand and sign a study-specific written informed consent prior to study entry.
* Patients receiving systemic therapy are eligible for this study if given >14 days prior to study entry and given no sooner than >14 days post radiation therapy (RT) completion.
* Complete history and general physical examination within 28 days prior to study entry

Exclusion Criteria:

* Known hypersensitivity to bendamustine or mannitol
* Patients with cerebral metastases from unknown primary tumors
* Patients with cerebral metastases from leukemias or lymphomas
* Patients with uncontrolled systemic cancer (i.e. evidence of systemic disease progression < 3 months prior to study entry)
* Systemic chemotherapy ≤14 days prior to study entry or ≤14 days after completing radiotherapy
* Patients who received prior BCNU wafer (Gliadel®) implantation for surgically resected cerebral metastatic lesions
* Patients with a life expectancy of less than 3 months
* Patients who received prior whole brain radiation therapy. As noted above, patients who received prior radiosurgery are allowed
* Patients with significant hydrocephalous
* Active clinically serious infection > Common Terminology Criteria for Adverse Events (CTCAE) Grade 2
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 24 Weeks per Patient
  To determine the MTD of bendamustine in combination with WBRT

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | 24 Weeks per Patient
  To determine the toxicity profile of bendamustine in combination with WBRT

CONTACTS AND LOCATIONS:
Overall Officials: Edward Pan, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States